CLINICAL TRIAL: NCT01683227
Title: Screening and Brief Intervention for Latino and Non-Latino White Drug Users
Brief Title: Screening, Brief Intervention, and Referral to Treatment for Drug Use
Acronym: SBIRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Susan I. Woodruff, Professor, San Diego State University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 1RC1DA028031-01 (NIH)
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Drug Abuse
Keywords: drug use; emergency department; brief intervention
MeSH Terms: conditions — Substance-Related Disorders; Emergencies | interventions — Mass Screening

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Screening/motivational drug intervention (Experimental): Screening and brief intervention counseling matched to patient's risk level delivered in the ER
  Interventions: Behavioral: Screening/motivational drug intervention
- Motivational placebo intervention (Placebo Comparator): Screening and brief intervention for driving and traffic safety
  Interventions: Behavioral: Motivational placebo intervention

INTERVENTIONS:
Behavioral: Screening/motivational drug intervention — Screening and brief motivational intervention delivered in the ER to reduce drug use
  Other Names: SBIRT
  Arms: Screening/motivational drug intervention
Behavioral: Motivational placebo intervention — Screening and brief motivational intervention delivered in the ER to reduce driving and traffic risk
  Arms: Motivational placebo intervention

SUMMARY:
Screening, Brief Intervention, and Referral to Treatment (SBIRT) is a comprehensive, integrated public health approach to identify and deliver a spectrum of early detection and intervention services for substance use in general medical care settings. These settings, such as emergency department visits, offer a potential "teachable moment" because patients may have perceptions of vulnerability about their health, and therefore be particularly receptive to screening and counseling. There is mounting scientific evidence suggesting SBIRT is effective in reducing alcohol use at varying levels of severity in a myriad of health care settings including primary care, emergency departments, and trauma centers. Although the SBIRT approach has shown promise for alcohol, relatively little is known about its effectiveness for adult illicit drug use specifically.

This will be among the first studies to rigorously test the SBIRT approach for drug use. It will evaluate the effectiveness of SBIRT for drug use and related factors for 700 multi-ethnic ED patients using a two-group randomized repeated-measures design in which biologically-validated drug use abstinence and related outcomes of an intervention group are compared to those of an attention-placebo control group. Over a 14-month period, bilingual/bicultural Health Educators recruited participants who reported past 30-day illicit drug use in excess of risky alcohol use from the waiting areas of two large hospital's ED and trauma units. Following consent procedures and standardized baseline assessments, Health Educators randomly assigned participants to one of the two conditions. The intervention group received "Life Shift," an SBIRT drug use intervention matched to the participant's drug use risk level. The control group received the same type and quantity of intervention in an unrelated area-Driving and Traffic Safety ("Shift Gears" program), also matched to their driving/traffic risk level. A 6-month face-to-face follow-up visit by trained measurement technicians blind to the participant's assigned condition collected standardized self-report past 30-day drug use measures (ASI-Lite)and hair samples for validating self-reported abstinence. Additional outcome variables are changes in the frequency of drug use, functional status measures (i.e., medical problems, psychiatric problems, and alcohol use), and health care utilization.

ELIGIBILITY:
Inclusion Criteria:

* 18 or over
* speak English or Spanish
* competent to give consent and interact
* drug use risk higher than alcohol use risk

Exclusion Criteria:

* under 18
* non english or spanish speaker
* no telephone where one can be reached
* too injured/sick to participate
* alcohol use risk higher than drug use risk

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
past 30 day drug use abstinence | 6 months post intervention
  Based on the addiction severity index-Lite

SECONDARY OUTCOMES:
Frequency of drug use | 6 months post intervention
  Based on composite score from the Addiction Severity Index-Lite

CONTACTS AND LOCATIONS:
Overall Officials: Susan I Woodruff, PhD, Principal Investigator — San Diego State University, School of Social Work
Locations (2):
- United States (2):
  - Scripps Mercy Emergency Department and Trauma Unit, San Diego, California
  - UCSD Emergency Department and Trauma Unit, San Diego, California

REFERENCES:
- [Derived] Woodruff SI, Clapp JD, Eisenberg K, McCabe C, Hohman M, Shillington AM, Sise CB, Castillo EM, Chan TC, Sise MJ, Gareri J. Randomized clinical trial of the effects of screening and brief intervention for illicit drug use: the Life Shift/Shift Gears study. Addict Sci Clin Pract. 2014 May 22;9(1):8. doi: 10.1186/1940-0640-9-8. PMID 24886786
- [Derived] Eisenberg K, Woodruff SI. Randomized controlled trial to evaluate screening and brief intervention for drug-using multiethnic emergency and trauma department patients. Addict Sci Clin Pract. 2013 Apr 8;8(1):8. doi: 10.1186/1940-0640-8-8. PMID 23566363